CLINICAL TRIAL: NCT06673745
Title: Comparative Effects of Instrument Assisted Soft Tissue Mobilisation and Dynamic Cupping on Elbow Range of Motion and Function in Children With Post Fracture Elbow Stiffness
Brief Title: Effect of Instrument Assisted Soft Tissue Mobilization and Dynamic Cupping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/24/0720
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Fractures, Bone
Keywords: elbow; post fracture stiffness
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: This will be a randomized clinical trail conducted on 28 participants of age 6 to 15 years .group A will get instrument assisted soft issue mobilisation and group B will get dynamic cupping therapy
Who Masked: Participant
Masking Description: This will be a randomized upping c clinical trial on 28 participant on 6 to 15 years group A will get instrument assisted soft tissue mobilisation and group B will get dynamic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrumental assisted soft tissue mobilization (Experimental): Instrument assisted soft tissue mobilization (IASTM) and dynamic cupping are manual therapy techniques used to address soft tissue restrictions and improve joint mobility and function. In the context of children with post-fracture elbow stiffness, these techniques can have several physiological effects. (14) This process involves the use of specialized tools to apply pressure and friction to the affected soft tissues. Which can help break down scar tissue and adhesions that may have formed following the fracture, allowing for improved tissue flexibility and mobility. This can stimulate blood flow to the area, promoting tissue healing and reducing inflammation
  Interventions: Other: IASTM
- Dynamic cupping therapy (Experimental): Dynamic cupping, on the other hand, utilizes suction cups placed on the skin to create negative pressure. This can help stretch and release tight muscles and fascia, increasing tissue flexibility and reducing stiffness. The rhythmic movement of the cups which can also stimulate lymphatic drainage and promote circulation, this will increase the removal of metabolic waste products and will also reduce swelling. (16) Both the techniques can help address the underlying soft tissue restrictions and joint stiffness commonly seen following a fracture. By improving tissue flexibility reducing inflammation, and enhancing circulation IASTM and dynamic cupping can contribute to restoring normal elbow range of motion and function in children with post fracture elbow stiffness. Instrument assisted soft tissue mobilization is one of the recently used popular myofascial intervention. It is known to improve the range of motion, function and improvestrigger point of the muscles. In recent studies it i
  Interventions: Other: Dynamic cupping therapy

INTERVENTIONS:
Other: IASTM — Group A received IASTM treatment, which will be given by the "Edge tool", that is an ergonomically designed stainless steel instrument and offers several different hand holds, eliminating operator fatigue. Prior to the treatment, the IASTM therapeutic effects will be explained. The scanning assessment will be done to identify areas of restrictions directed by the gritty sensations using the Edge tool. Each restriction will be treated with the tool for 30-60 sec and given. This treatment will be given for 30 minutes for 3 days per week for 4 weeks
  Arms: Instrumental assisted soft tissue mobilization
Other: Dynamic cupping therapy — On the contrary, group B the patient will be seated in a chair with the elbow flexed on the plinth to relax the forearm muscles. The area around the elbow joint will be cleaned with alcohol to remove any foreign bodies from the treated area. Dynamic cupping therapy for elbow stiffness will begin with an assessment of the patient's condition, where factors such as the extent of stiffness and range of motion in the elbow joint will be evaluated. Following this assessment, lubricant will be applied to the skin surrounding the elbow to facilitate smooth movement of the cups. Cups of suitable size and material will then be strategically placed around the elbow joint, and suction will be created inside each cup to create a vacuum effect. Once thesecurely attached, the practitioner will move them around the elbow area using gentle techniques such as gliding or pumping motions.
  Arms: Dynamic cupping therapy

SUMMARY:
Children who experience fractures may develop stiffness and limited range of motion in their affected joints, notably the elbow. Although conventional rehabilitation approaches have demonstrated some effectiveness, innovative methods like Instrument Assisted Soft Tissue Mobilization (IASTM) and Dynamic Cupping hold promise for enhancing outcomes. These techniques represent emerging therapies aimed at improving range of motion and function across different musculoskeletal conditions. However, there is a lack of comparative research examining their efficacy specifically in pediatric patients with post-fracture elbow stiffness

DETAILED DESCRIPTION:
This will be a randomized clinical trial conducted on 28 participants. Data will be collected from Khatoon e Jannat hospital, Mujahid hospital and children hospital of Faisalabad. The study includes children aged 6 to 15, both genders, experiencing elbow postoperative stiffness and with a loss of extension of at least -30 degrees and/or flexion of no more than 120 degrees. Participants excluded from the study are those who declined consent, had pathological fractures, and associated ipsilateral injuries, bilateral upper extremity injuries, neuro-vascular disorders, heterotrophic ossification, or contraindications for IASTM. A sample of 28 will be divided in to two groups. Each group will consist of 14 participants. Group A will receive instrument assisted soft tissue mobilization. On the contrary group B will receive dynamic cupping therapy. Both groups will be given conventional therapy along with prescribed intervention. Intervention will be given for 30 minutes for 3 sessions per week for 4 weeks. Data will be collected before and after the intervention to assess range of motion and function with a help of goniometer and Disability arm shoulder and hand questionnaire. Data will be analyzed by using SPSS version 26.0

ELIGIBILITY:
Inclusion criteria

* Age from 6 to 15 years (23)
* Both genders Participant with elbow postoperative stiffness with loss of extension of ≥-30 degrees and/or flexion ≤120 degrees Participant with at least 6-week post-surgery with open reduction and internal fixation done for either of the following fractures.

Exclusion Criteria:

* Participants who declined consent.
* Participants who had pathological fractures, associated ipsilateral injuries, bilateral upper extremity injuries, neuro-vascular disorders, heterotrophic ossification, and contraindications for IASTM

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand Questionnaire | 6 weeks
  Function was assessed by the Disability of arm shoulder and hand questionnaire (DASH) (Reliability- ICC- 0.96; validity- 0.70), which is a 30-item patient-reported questionnaire, which can rate difficulty and interference with function on a 5-point Likert scale used to evaluate impairments, activity limitations, as well as participation restrictions in both leisure activities and work due to elbow dysfunction, regardless of which arm is affected. The scores for all items are then summed up to a scale score, where higher scores indicate higher disability
Goniometer Measurement for Range of motion | 6 weeks
  Universal goniometer is a device which is used to measure the range of motion of the joint. It has both art and science of measuring joint plane by 2 form. It has short and long arm. It has 3 parts Center part is known as fulcrum or axis with two arms. One is moving arm and the other is stationary or fixed arm. ROM of the elbow joint and forearm was measured using the universal half goniometer (Reliability-ICC-0.53-0.97.) Positions used to measure elbow flexion-extension were in supine position, whereas the forearm pronation-supination was done in sitting position .
Numeric Pain rating Scale | 6 weeks
  Numeric pain rating scale is a subjective measure 11 point numerical scale which is used to measure pain. Is scoring range In this scale 0 shows no pain and 10 shows worst pain imaginable. It has good reliability of 0.79 and validity of 0.96. (26)

CONTACTS AND LOCATIONS:
Overall Officials: Sana Aziz, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Instrument assisted soft tissue mobilization (IASTM) and dynamic cupping are manual therapy techniques used to address soft tissue restrictions and improve joint mobility and function. In the context of children with post-fracture elbow stiffness, these techniques can have several physiological effects. (14) This process involves the use of specialized tools to apply pressure and friction to the affected soft tissues. Which can help break down scar tissue and adhesions that may have formed following the fracture, allowing for improved tissue flexibility and mobility. This can stimulate blood flow to the area, promoting tissue healing and reducing inflammation. (15) Dynamic cupping, on the other hand, utilizes suction cups placed on the skin to create negative pressure. This can help stretch and release tight muscles and fascia, increasing tissue flexibility and reducing stiffness. The rhythmic movement of the cups which can also stimulate lymphatic drainage and promote circulation, thi

REFERENCES:
- [Background] Aksan Sadikoglu B, Analay Akbaba Y, Taskiran H. Effects of ischemic compression and instrument-assisted soft tissue mobilization techniques in trigger point therapy in patients with rotator cuff pathology: randomized controlled study. Somatosens Mot Res. 2022 Mar;39(1):70-80. doi: 10.1080/08990220.2021.2005015. Epub 2021 Nov 24. PMID 34818976